CLINICAL TRIAL: NCT05426824
Title: A Prospective, Multi-center Study of Whole-course Management of Pegaspargase in Extranodal NK/T Cell Lymphoma (ENKTL)
Brief Title: The Whole-course Management of Pegaspargase in ENKTL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-SR-059
Record Dates: First submitted 2022-03-31; First posted 2022-06-22 (Actual); Last update posted 2022-06-22 (Actual); Status verified 2022-06

CONDITIONS: Extranodal NK/T Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P-GOD (Experimental): P-GOD (peasparaginase + gemcitabine + oxaliplatin + dexamethasone) ;
  Interventions: Drug: Pegaspargase（P-GOD）
- PEMD (Experimental): PEMD (peaspargase + etocytidine + methotrexate + dexamethasone)
  Interventions: Drug: Pegaspargase（PEMD）

INTERVENTIONS:
Drug: Pegaspargase（P-GOD） — stage I/II) ENKTL patients receiving P-GOD for the first time, gemcitabine 1000 mg/m2 intravenously on day 1 and day 5, oxaliplatin 75 mg/m2 intravenously on day 1, dexamethason 40 mg intravenously on day 1-4, and pegaspargase 3750 IU intramuscularly on day 2. The cycle was repeated every 21 days.The activity of pegaspargase in peripheral blood will be detected on D3, D4, D5, D6, D7, D8, D10, D12, D14, D16, D18 and D21.
  Arms: P-GOD
Drug: Pegaspargase（PEMD） — stage III/IV ENKTL patients receiving PEMD for the first time,methotrexate 3.0 g/m2 intravenously over 6 h on day 1, etoposide 100 mg/m2 intravenously on days 2-4, dexamethasone 40 mg intravenously on days 1-4, pegaspargase 3750 IU intramuscularly on day 2. The activity of pegaspargase in peripheral blood will be detected on D3, D4, D5, D6, D7, D8, D10, D12, D14, D16, D18 and D21.
  Arms: PEMD

SUMMARY:
This is a prospective, multi-center study of the whole-course management of pegaspargase in Extranodal NK/T cell lymphoma (ENKTL). Based on a complete population pharmacokinetic model of pegaspargase in ENKTL patients, the time node of asparaginase monitoring and the principle of dose adjustment will be formulated. Besides, the proportion of "silent inactivation" of asparaginase in ENKTL patients and its effect on the prognosis of patients will also be explored. The treatment plan is as follows: (1) During 8 early (stage I/II) ENKTL patients receiving P-GOD (peasparaginase + gemcitabine + oxaliplatin + dexamethasone) for the first time, the activity of pegaspargase in peripheral blood will be detected on D3, D4, D5, D6, D7, D8, D10, D12, D14, D16, D18 and D21. (2) During 4 early (stage III/IV) ENKTL patients receiving PEMD (peaspargase + etocytidine + methotrexate + dexamethasone) for the first time, the activity of pegaspargase in peripheral blood will be detected on D3, D4, D5, D6, D7, D8, D10, D12, D14, D16, D18 and D21. (3) During 72 (including above 12 patients) ENKTL patients receiving P-GOD/PEMD, the activity of pegaspargase and anti-pegaspargase in peripheral blood will be detected on D9 and D16 of each cycle of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed first-line ENKTL patients according to WHO 2016
* Willingness to provide written informed consent.

Exclusion Criteria:

* Patients are unsuitable for the enrollment according to investigator's judgement.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2024-07-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Plasma activity curve of pegaspargase | Plasma activity measurement of pegaspargase [time frame: Day3, Day4, Day5, Day6, Day7, Day8, Day10, Day12, Day14, Day16, Day18, and Day21 of first use of pegaspargase]
  pegaspargase in ENKTL patients

SECONDARY OUTCOMES:
the proportion of "silent inactivation" | days 7, 14, 21 of treatment
  asparaginase in ENKTL patients

OTHER OUTCOMES:
The 2-year PFS rate | 2-year of Treatment
AUC | Days 7, 14 of treatment
MIC | Days 7, 14 of treatment (steady state)
Cmax | Days 7, 14 of treatment (steady state)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, Principal Investigator — The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital)
Locations (1):
- Hematological Department, People's Hospital of Jiangsu Province, Nanjing, Jiangsu, China